CLINICAL TRIAL: NCT03783910
Title: Cross-over Multiple Dose Study Assessing the Analgesic Efficacy and Safety of Oral GRT9906 Compared to Placebo in Subjects With Primary Fibromyalgia Syndrome
Brief Title: Efficacy and Safety of GRT9906 Tablets Compared to Placebo in Patients With Fibromyalgia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF9906/03
Record Dates: First submitted 2018-12-18; First posted 2018-12-21 (Actual); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Primary Fibromyalgia
Keywords: Chronic pain
MeSH Terms: conditions — Fibromyalgia; Chronic Pain | interventions — 3-(2-dimethylaminomethylcyclohexyl)phenol

STUDY DESIGN:
Intervention Model Description: This dose-titration study was conducted with randomized, multi-center, double-blind, placebo-controlled, crossover design and multiple administrations in 2 treatment sequences in treatment periods 1 and 2: Sequence GRT9906-Placebo and sequence Placebo-GRT9906.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GRT9906 (Experimental): Participants received 80-240 mg of GRT9906 oral for up to 6 weeks (1 week of titration, 5 weeks of maintenance treatment).
  Participants started with 40 mg of GRT9906 on the first and 80 mg (40 mg twice daily) on the second day. They could increase the dose every day by 1 tablet (i.e., GRT9906 40 mg), up to a maximum daily dose of 240 mg (120 mg twice daily). Participants experiencing adverse events could reduce the dose to the next lower, better tolerated daily dose (but not lower than 80 mg [40 mg twice daily]). By Day 8, every participant had reached their optimal daily dose and was asked to continue on the identified dosing regimen for the following 5 weeks.
  Interventions: Drug: GRT9906
- Placebo (Placebo Comparator): Participants received Placebo (2-6 tablets daily) oral for up to 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GRT9906 — One prolonged-release tablet containing 40 mg of GRT9906
  Arms: GRT9906
Drug: Placebo — Placebo matching GRT9906 tablets
  Arms: Placebo

SUMMARY:
The study was performed in participants suffering from fibromyalgia and investigated efficacy after treatment with several doses of GRT9906 versus placebo. Furthermore, it was to be found out if treatment with GRT9906 was safe and well-tolerated.

DETAILED DESCRIPTION:
This Phase 2 study had a randomized, multi-center, double-blind, placebo-controlled, crossover, multiple-administration design.

The objectives of the study were the following:

* To assess the multiple-dose analgesic efficacy and safety of an oral prolonged-release (PR) tablet formulation of GRT9906 at daily doses between 80 and 240 milligrams (mg) in comparison to placebo in participants with moderate to severe pain due to primary fibromyalgia syndrome (FMS).
* To compare the tolerability of multiple-dose GRT9906 PR to placebo in participants with primary FMS.
* To generate data that could be used, in combination with data from other studies, to explore the population pharmacokinetic analysis and pharmacokinetic/pharmacodynamic (PK/PD) properties of GRT9906 PR.

The study consisted of 5 phases:

1. Enrollment including tapering, if necessary, and washout (at least 1 week) of previous medication.
2. First treatment period with 1-week titration and 5-weeks dosing on participant's last well-tolerated titration dosage.
3. Interim washout period of at least 1 week.
4. Second treatment period with 1-week titration and 5-weeks dosing on participant's last well-tolerated titration dosage.
5. Final washout period of at least 1 week, terminated by a Follow-up Visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ambulatory participants of any ethnic group, aged 18 to 75 years inclusive at enrollment.
* Primary fibromyalgia syndrome (FMS) diagnosed according to the American College of Rheumatology (ACR) 1990 criteria, persistent for at least 6 months.
* Average Pain Intensity of FMS pain over the last 3 days before randomization visit must be at least 4 points, using 11-point numerical rating scale (NRS).
* Negative urine test for drugs of abuse at the Day 1 visit of each treatment period.
* Women of childbearing potential must use an acceptable method of contraception (i.e., double barrier, hormonal or intra-uterine device method) during the study period and have a negative urine pregnancy test at the Enrollment Visit and at the Day 1 visit of each treatment period.
* Compliance with use and completion of assessments by means of electronic diaries; 80 percent of entries must be available for the week before randomization.
* Written informed consent for study participation given.

Exclusion Criteria:

* Participation in another study of IMPs or devices parallel to, or less than 1 month prior to enrollment, or previous participation in this study.
* Known to or suspected of not being able to comply with the study protocol and the use of the IMPs.
* Not able to communicate meaningfully with the Investigator and staff.
* Evidence or history of alcohol, medication or drug dependency during the past 12 months. History of opiate dependency at any point in life.
* Evidence or history of neurotic personality, psychiatric illness including anxiety disorder, severe senile dementia, Alzheimer's disease, history of seizures or pre-existing conditions that lower seizure threshold (e.g., head trauma), or suicide risk.
* Current depression needing treatment with antidepressants.
* Currently or previously diagnosed with malignancies except basal cell carcinoma; poor medical status (e.g., New York Heart Association [NYHA] class equal to or above 3; Child classification for hepatic impairment above A [Pugh et al. 1973]; decompensated chronic obstructive pulmonary disease) or, at the discretion of the Investigator, clinical signs that raise concerns about participant's suitability for the study.
* Creatinine higher than 1.5-times of upper limit of normal (ULN) range.
* Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) higher than twice the ULN range.
* Any chronic disease (e.g., hepatic, renal and/or gastrointestinal) that might affect drug absorption, metabolism or excretion.
* Nursing mother.
* Causes of chronic pain other than FMS and mild osteoarthritis of the hand.
* Proven rheumatoid disease with positive rheumatoid factor or antinuclear antibody (ANA) at screening.
* History of marked repolarization abnormality (e.g., suspicion of or definite congenital long QT syndrome).
* QT values of: corrected QT Bazett (QTcB) females equal to or above 450 milliseconds (ms), QTcB males equal to or above 430 ms, uncorrected QT equal to or above 500 ms at Enrollment Visit.
* Definite or suspected allergy or hypersensitivity to drugs having a similar mechanism of action as IMP. Known contraindications/hyper-sensitivity to opioids, acetaminophen or zolpidem.
* Intolerance to galactose.
* Dysphagia or difficulty swallowing tablets or capsules.
* Blood donation (above 100 milliliters) or comparable blood losses within 3 months prior to the start of this study.
* History of Gilbert's Disease.
* Use of anti-epileptic drugs, chloramphenicol, rifampicin, or zidovudine.
* Use of fentanyl transdermal system, buprenorphine sublingual or transdermal system, cyclooxygenase (COX) 2 inhibitors with a half-life of more than 35 hours, equal to or less than 7 days prior to enrollment.
* Use of serotonergic drugs, drugs with the potential to prolong QT interval, cytochrome P450, family 2, subfamily D, polypeptide 6 (CYP2D6) substrates, antiparkinson drugs, monoamineoxidase (MAO)-inhibitors, neuroleptics, or other drugs that may lower the seizure threshold, within less than 5 half-life times prior to randomization.
* Use of any analgesics (including non-steroidal anti-inflammatory drugs [NSAIDs] and COX2 inhibitors) others than investigational medicinal products and acetaminophen as rescue medication as well as sedative hypnotics (with the exception of 5 milligrams zolpidem for a maximum of 3 days per week) within less than 5 half-life times prior to randomization.
* Physical therapy and/or other non-pharmacological pain therapy (e.g., acupuncture, transcutaneous electrical nerve stimulation [TENS]) after Enrollment Visit if not started at least 6 months before enrollment.
* Systemic (parenteral and/or oral) steroids during previous month.
* Tender point injections (with local anesthetics or others) during the previous month.
* Participants currently involved in litigation regarding FMS, pending or active disability-compensation claim.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2005-09-19 (Actual); Primary Completion 2006-10 (Actual); Study Completion 2006-10-20 (Actual)

PRIMARY OUTCOMES:
Average Pain Intensity over last 3 days of treatment period | Last 3 days of treatment period
  Participants recorded their daily current pain intensity in an electronic diary from the Enrollment Visit until the day of the last visit in the second treatment period using an 11-point Numerical Rating scale (NRS) ranging from 0 = no pain to 10 = pain as bad as you can imagine. Each treatment period lasted for 6 weeks. For the primary endpoint, the average daily current pain intensity over the last 3 days prior to the last visit per treatment period was calculated.

SECONDARY OUTCOMES:
Changes from baseline/period baseline in Average Pain Intensity over last 3 days per treatment period | At baseline, at period baseline, and for last 3 days of each treatment period
  Participants recorded their daily current pain intensity in an electronic diary from the Enrollment Visit until the day of the last visit in the second treatment period using an 11-point Numerical Rating scale (NRS) ranging from 0 = no pain to 10 = pain as bad as you can imagine. Each treatment period lasted for 6 weeks. Changes from baseline/period baseline for the average daily current pain intensity over the last 3 days prior to the last visit per treatment period were calculated.
Average Pain Intensity after initial washout and over Weeks 1 to 6 per treatment period | Last 3 days of the initial washout period; Week 1, 2, 3, 4, 5 and 6 per treatment period
  Participants recorded their daily current pain intensity in an electronic diary from the Enrollment Visit until the day of the last visit in the second treatment period using an 11-point Numerical Rating scale (NRS) ranging from 0 = no pain to 10 = pain as bad as you can imagine. Each treatment period lasted for 6 weeks. The average daily current pain intensities over the last 3 days of the initial washout period (before randomization) and over Weeks 1, 2, 3, 4, 5, and 6 per treatment period were calculated.
Fibromyalgia Impact Questionnaire (FIQ) | At Enrollment Visit (Visit 1), on Day 1, Day 22, and Day 42 per treatment period, and at Final Visit (14 days after last dose in treatment period 2)
  The FIQ is a 10-item self-administered questionnaire measuring physical functioning, work status, depression, anxiety, sleep, pain, stiffness, fatigue, and well-being over a 1-week period. Each of the 10 items has a maximum possible score of 10 with a higher score indicating a greater impact of the syndrome on the patient. The FIQ total score is calculated by a weighted sum of the 10 items. The FIQ total score and sub-scores for FIQ items for fatigue, tiredness on awakening, and stiffness were calculated.
Tender Point Index (TPI) | At Enrollment Visit (Visit 1), on Day 1, Day 22, and Day 42 per treatment period, and at Final Visit (14 days after last dose in treatment period 2)
  Digital palpation with an approximate force of 4 kg was applied at 18 tender point sites. A tenderness scale was applied to the tenderness at each tender point site examined: non-tender (0), tender without physical response (1), tender plus wince or withdrawal (2), exaggerated withdrawal (3), too painful to touch (4). The sum of the tenderness severities at all 18 sites was the TPI. The expected range for normal controls is 0-5, for participants with fibromyalgia 11-72.
Average Pain Threshold (APT) | At Enrollment Visit (Visit 1), on Day 1, Day 22, and Day 42 per treatment period, and at Final Visit (14 days after last dose in treatment period 2)
  A Fischer algometer was used for this purpose. The foot piece was placed on the skin at the site of each tender point. The axis of the instrument was held firmly in place by a finger or thumb and vertical to the skin surface. The participant was informed that they "will at first feel only pressure but then it will change to pain". The participant was to say "now" at the exact time when the pressure feeling changed to a pain feeling. The algometer applied pressure was advanced at a rate of 1 kg/second. When the participant indicated "now" the examiner withdrew the instrument and read the gauge pressure in kg to one decimal place. A value was recorded for algometry at each of the 18 tender points. The average of these 18 values has been defined as the APT.
Morning Stiffness Questionnaire (MSQ) | At Enrollment Visit (Visit 1), on Day 1, Day 22, and Day 42 per treatment period, and at Final Visit (14 days after last dose in treatment period 2)
  The duration of morning stiffness during the past 7 days was assessed by answering 3 questions, each with 5 categories of "no stiffness" and "1 hour", "2 hours", "3 hours", or "5 hours". Questions were "During the past 7 days, on average, how long did your morning stiffness last until it began to improve/maximum improvement occurred/how long did it take to get going properly?".
Major Depression Inventory (MDI) | At Enrollment Visit (Visit 1), on Day 1, Day 22, and Day 42 per treatment period, and at Final Visit (14 days after last dose in treatment period 2)
  The MDI scale is a 10-item self-administered questionnaire for assessing major depression according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) and International Classification of Diseases (ICD-10) as well as measuring severity of depressive states. Each item is scored on a Likert scale from 0 to 5. Treatment outcome is measured by the sum of the 10 individual items. In addition to the total score, a MDI rating scale was defined as follows: No sign of Depression: MDI total score below 20; Mild Depression: MDI total score of 20 to 24; Moderate Depression: MDI total score of 25 to 29; Severe Depression: MDI total score of 30 and more.
Change from baseline in Sleep Problem Scale (SPS) total score | At Enrollment Visit (Visit 1) and on Day 42 per treatment period
  The SPS is a 4-item questionnaire assessing sleep problems over a 1-month period, covering the following dimensions: delay of sleep onset, difficulty staying asleep, awakening too early, and tiredness after usual amount of sleep. Response categories comprised: Not at all (score 0), 1-3 days (1), 4-7 days (2), 8-14 days (3), 15-21 days (4), and 22-31 days (5). The SPS total score is calculated as the sum of the 4 individual items. Greater levels of sleep problems are indicated by higher scores. The SPS total score is calculated as the sum of the 4 individual items. Changes from baseline (Visit 1) for the SPS total score at Day 42 are calculated per treatment period.
30 percent reduction in pain based on Average Pain Intensity (API) | Prior to the last visit in each treatment period (Day 42)
  The number of participants who achieved a 30 percent reduction in pain is calculated based on the API recorded prior to the last visit in each treatment period. The dichotomous variable (yes/no) is calculated separately for each period. A participant with at least a 30 percent reduction in pain from period/overall baseline is coded as 30 percent reduction = Yes.
50 percent reduction in pain based on Average Pain Intensity (API) | Prior to the last visit in each treatment period (Day 42)
  The number of participants who achieved a 50 percent reduction in pain is calculated based on the API recorded prior to the last visit in each treatment period. The dichotomous variable (yes/no) is calculated separately for each period. A participant with at least a 50 percent reduction in pain from period/overall baseline is coded as 50 percent reduction = Yes.
Number needed to treat (NNT) for 30 percent reduction in pain | Prior to the last visit in each treatment period (Day 42)
  The number of participants needed to be treated with GRT9906 to achieve 1 additional participant with a 30 percent reduction in pain prior to the last visit in each treatment period was calculated based on the number of participants with a 30 percent reduction in API values.
Number needed to treat (NNT) for 50 percent reduction in pain | Prior to the last visit in each treatment period (Day 42)
  The number of participants needed to be treated with GRT9906 to achieve 1 additional participant with a 50 percent reduction in pain prior to the last visit in each treatment period was calculated based on the number of participants with a 50 percent reduction in API values.
Quality of sleep using the Sleep Problem Scale (SPS) | At Visit 1 and on Day 42 of each treatment period
  The SPS total score is calculated as the sum of the 4 individual items. Change will be calculated by subtracting the SPS total score obtained at baseline (Visit 1) from the SPS total score obtained at Day 42 per treatment period.
Subject's Global Assessment of the investigational medicinal product (IMP) | On Day 42 of each treatment period
  The participant rated their overall impression of the IMP at Day 42 or final visit per treatment period. They were asked the following questions on a 5-point verbal rating scale (VRS): "How would you rate the IMP you received for pain?" Excellent (4), Very Good (3), Good (2), Fair (1), Poor (0). Frequencies per category were calculated.
Investigator's Global Assessment of the investigational medicinal product (IMP) | On Day 42 of each treatment period
  Physicians rated their overall impression of the IMP at Day 42 or final visit per treatment period. They were asked the following questions on a 5-point VRS: "How would you rate the IMP the subject received for pain?" Categories were Excellent (4), Very Good (3), Good (2), Fair (1), Poor (0). Frequencies per category were calculated.
Patient's Global Impression of Change (PGIC) | On Day 42 of each treatment period
  Participants rated their overall impression of change on a 7-point VRS: "Compared to your pain at admission to the project, how much has it changed?" Categorical scales are: Very much improved (1), Much improved (2), Minimally improved (3), No change (4), Minimally worse (5), Much worse (6), Very much worse (7). Frequencies per category are calculated.
Mean daily number of rescue medication tablets taken | From Day 1 to Day 42 over each treatment period
  Rescue medication (acetaminophen up to 2 grams per day) was allowed in the study. The mean daily amount (mg/day) was determined per treatment period.
Total amount of rescue medication taken | From Day 1 to Day 42 over each treatment period
  Rescue medication (acetaminophen up to 2 grams per day) was allowed in the study. The total amount (mg) was determined per treatment period.
Clinical Opiate Withdrawal Scale (COWS) | At Visit 1 and Day 45 (2-4 days after last day of intake of IMP per treatment period)
  Withdrawal symptoms were assessed using the COWS questionnaire. It comprises 11 items (resting pulse while sitting or lying for 1 minute, gastrointestinal upset over last half hour, sweating over past half hour, tremor observed with outstretched hands, restlessness during assessment, yawning during assessment, pupil size, anxiety or irritability, bone or joint aches attributed to opiate withdrawal, gooseflesh skin, runny nose or tearing not accounted for by cold symptoms or allergies) that best describe the participants' signs or symptoms. Point values of each answer to be included in the total score vary between 0 and 5 (the higher the value the worse). The sum of all 11 items is rated as follows: 5-12 = mild, 13-24 = moderate, 25-36 = moderately severe, above 36 = severe withdrawal.

CONTACTS AND LOCATIONS:
Overall Officials: Grünenthal Study Director, Study Director — Grünenthal GmbH
Locations (6):
- United States (6):
  - 006 Research Facility, DeLand, Florida
  - 005 Research Facility, Charlotte, North Carolina
  - 004 Research Facility, Medford, Oregon
  - 002 Research Facility, Portland, Oregon
  - 001 Research Facility, San Antonio, Texas
  - 003 Research Facility, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pugh RN, Murray-Lyon IM, Dawson JL, Pietroni MC, Williams R. Transection of the oesophagus for bleeding oesophageal varices. Br J Surg. 1973 Aug;60(8):646-9. doi: 10.1002/bjs.1800600817. No abstract available. PMID 4541913